CLINICAL TRIAL: NCT04537806
Title: A Study of Brexanolone for Acute Respiratory Distress Syndrome Due to COVID-19
Brief Title: A Study of Brexanolone for Acute Respiratory Distress Syndrome (ARDS) Due to Coronavirus Disease 2019 (COVID-19)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Internal company decision
Sponsor: Sage Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 547-ARD-301
Record Dates: First submitted 2020-09-01; First posted 2020-09-03 (Actual); Results first posted 2022-07-27 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19 | interventions — brexanolone; Pregnanolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants receiving mechanical ventilation as standard of care were randomized to receive a 60-hour single continuous intravenous (IV) infusion of brexanolone-matching placebo.
  Interventions: Drug: Placebo
- Brexanolone (Experimental): Participants receiving mechanical ventilation as standard of care were randomized to receive a 60-hour single continuous IV infusion of brexanolone at 70 micrograms per kilogram per hour (mcg/kg/h) for 58 hours followed by a 2-hour taper of brexanolone at 35 mcg/kg/h.
  Interventions: Drug: Brexanolone

INTERVENTIONS:
Drug: Brexanolone — Administered as IV infusion.
  Other Names: Allopregnanolone; Zulresso; SAGE-547
  Arms: Brexanolone
Drug: Placebo — Administered as IV infusion.
  Arms: Placebo

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of brexanolone in participants on ventilator support for acute respiratory distress syndrome (ARDS) due to COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Participant was confirmed positive for the novel coronavirus responsible for SARS-CoV-2 (severe acute respiratory syndrome coronavirus 2) infection as determined by polymerase chain reaction (PCR) at Screening
* Participant had a presumptive diagnosis of ARDS at Screening and partial pressure of arterial oxygen (PaO2)/fraction of inspired oxygen (FiO2) (ratio of partial pressure of arterial oxygen to fraction of inspired oxygen [PF ratio]) less than (<) 300 prior to randomization
* Participant was intubated and receiving mechanical ventilation prior to randomization
* Participants must had initiated mechanical ventilation within 48 hours prior to screening, or had an immediate clinical plan for such intervention at time of screening
* Participant was likely to survive, in the opinion of the investigator, for at least 72 hours from the time of screening

Exclusion Criteria:

* Participant had fulminant hepatic failure at Screening
* Participant had end stage renal disease at Screening
* Participant had a known allergy to progesterone, allopregnanolone, or any excipients in the brexanolone injection
* Participant was concurrently participating in another clinical trial for an investigational product or device at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-12-18 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Sage Investigational Site, Fresno, California
  - Sage Investigational Site, Augusta, Georgia
  - Sage Investigational Site, Boston, Massachusetts
  - Sage Investigational Site, Burlington, Massachusetts
  - Sage Investigational Site, Lansing, Michigan
  - Sage Investigational Site, Las Vegas, Nevada
  - Sage Investigational Site, Charlotte, North Carolina
  - Sage Investigational Site, Richmond, Virginia
  - Sage Investigational Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Data sharing will be consistent with the results submission policy of ClinicalTrials.gov.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in the study at 9 centers in the United States from 18 December 2020 to 01 July 2021.
Pre-assignment Details: A total of 33 participants were screened of which 29 were randomized and 28 were dosed. This study consisted of up to a 2-day screening period, a 60-hour treatment period plus an additional follow-up of up to 23 days.
Period: Overall Study
Arm/Group | Placebo | Brexanolone
Started | 15 | 14
Safety Analysis Set (Safety analysis set included all participants who initiated Investigational product (IP) (brexanolone or placebo).) | 14 | 14
Full Analysis Set (Full analysis set (FAS) included all randomized participants who initiated IP (brexanolone or placebo).) | 14 | 14
Completed | 13 | 13
Not Completed | 2 | 1
Not completed — Randomized but not treated | 1 | 0
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Population: FAS included all randomized participants who initiated IP (brexanolone or placebo).
Groups:
- Placebo: Participants receiving mechanical ventilation as standard of care were randomized to receive a 60-hour single continuous IV infusion of brexanolone-matching placebo.
- Brexanolone: Participants receiving mechanical ventilation as standard of care were randomized to receive a 60-hour single continuous IV infusion of brexanolone at 70 mcg/kg/h for 58 hours followed by a 2-hour taper of brexanolone at 35 mcg/kg/h.
- Total: Total of all reporting groups
Arm/Group | Placebo | Brexanolone | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.6 (9.81) | 58.2 (12.79) | 60.4 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 14
  Male | 8 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 11 | 10 | 21
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 1 | 2
  Race: Black or African American | 2 | 1 | 3
  Race: White | 10 | 11 | 21
  Race: Other | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Alive and Free of Respiratory Failure at Day 28
Description: Respiratory failure is defined based on resource utilization, requiring at least one of the following: Endotracheal intubation and mechanical ventilation, oxygen delivered by high-flow nasal cannula (heated, humidified oxygen delivered via reinforced nasal cannula at flow rates >20 liter/minute with fraction of delivered oxygen >=0.5), noninvasive positive pressure ventilation, and extracorporeal membrane oxygenation (ECMO). Percentage of participants who were alive and free of respiratory failure at Day 28 were reported in this outcome measure.
Time Frame: Day 28
Population: FAS included all randomized participants who initiated IP (brexanolone or placebo). Here, "Overall number of participants analyzed" signifies the number of participants with available data for analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brexanolone
Number analyzed (Participants) | 13 | 13
percentage of participants | 23.1 | 23.1
Statistical Analysis 1: Comparison: Placebo vs Brexanolone; Test type: Superiority; p = 1.0000, Chi-squared; Proc Genmod = 0.0, 95% CI 2-sided [-31.8 to 31.8] — Estimates for treatment, and the corresponding 95% confidence interval (CI) were estimated using Proc Genmod method, with treatment as a factor and age groups as a covariate variable

2. Secondary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant administered with a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom or disease temporally associated with the use of an IP whether or not related to the product. An AE can include any undesirable medical condition, even if no study treatment has been administered. A TEAE is defined as an AE with onset after the start of IP, or any worsening of a pre-existing medical condition/AE with onset after the start of IP and throughout the study.
Time Frame: From first dose of investigational product up to end of study (up to Day 40)
Population: Safety analysis set included all participants who initiated IP (brexanolone or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brexanolone
Number analyzed (Participants) | 14 | 14
Participants | 13 | 14

3. Secondary Outcome: Number of Participants Who Died Through Day 28
Description: All cause mortality was reported up to Day 28 in this outcome measure.
Time Frame: From screening up to Day 28
Population: Safety analysis set included all participants who initiated IP (brexanolone or placebo).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brexanolone
Number analyzed (Participants) | 14 | 14
Participants | 6 | 8

ADVERSE EVENTS:
Time Frame: From screening up to end of study (up to Day 40)
Description: Safety analysis set included all participants who initiated IP (brexanolone or placebo).
Arm/Group | Placebo | Brexanolone
All-Cause Mortality (participants affected / at risk) | 7/14 | 8/14
Serious Adverse Events (participants affected / at risk) | 8/14 | 8/14
Other Adverse Events (participants affected / at risk) | 11/14 | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Brexanolone (N=14)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 2
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1
Pneumonia serratia (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 1
Endotracheal intubation (Surgical and medical procedures) | 2 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=14) | Brexanolone (N=14)
Septic shock (Infections and infestations) | 0 | 4
Candida infection (Infections and infestations) | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Bacterial disease carrier (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 2
Haematochezia (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 1
Penis injury (Injury, poisoning and procedural complications) | 0 | 1
Product administration interrupted (Injury, poisoning and procedural complications) | 0 | 1
Scrotal injury (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Ear injury (Injury, poisoning and procedural complications) | 1 | 0
Mechanical ventilation complication (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Delirium (Psychiatric disorders) | 0 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Intensive care unit delirium (Psychiatric disorders) | 1 | 0
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Metabolic alkalosis (Metabolism and nutrition disorders) | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 3 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Defect conduction intraventricular (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 1
Hypothermia (General disorders) | 1 | 0
Staphylococcus test positive (Investigations) | 0 | 1
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Tracheostomy (Surgical and medical procedures) | 1 | 1
Endotracheal intubation (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
The study was terminated early due to sponsor's decision and there were no safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI can either be a party and subject to the same restrictions as the institution, or if not a party, the restrictions are described on the face of the contract (i.e., PI is a contractor of the institution; PI is part of a larger group of study personnel; institution has contracted with or otherwise bound all study personnel under confidentiality obligations and requirements to vest intellectual property to the institution).

DOCUMENTS (2):
  • Study Protocol (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/06/NCT04537806/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/06/NCT04537806/SAP_001.pdf